CLINICAL TRIAL: NCT04678973
Title: Effects of Brief, mHealth Self-Compassion Intervention on Internalized Weight Bias in Adults With Obesity: A Randomized Controlled Trial
Brief Title: Brief mHealth Self-Compassion Intervention on Internalized Weight Bias
Acronym: ruby
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-0033
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Obesity; Stigma, Social
Keywords: mindfulness; self-compassion; mhealth
MeSH Terms: conditions — Obesity; Social Stigma

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups: self-compassion intervention or wait-list control group.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention group will receive a 4 week program delivered via text message. Week 1 will include psychoeducation delivered via brief readings and video. Weeks 2-4 will include daily guided mindfulness practice focusing on self-compassion and weight and body image concerns.
  Interventions: Behavioral: Self-compassion mindfulness practice
- Wait-list control (No Intervention): Participants in the control group will receive no study content during the 4 week intervention period. They will receive access to intervention content (text messages, audio files) after completing end-of-treatment surveys 4 weeks after randomization.

INTERVENTIONS:
Behavioral: Self-compassion mindfulness practice — Guided Mindfulness Practice: Participants in the intervention group will receive compassion-based guided meditation audio recordings. Recordings will target self-compassion and body concerns simultaneously.
  Psychoeducation: Participants in the intervention group will receive psychoeducation delivered via daily PDF over days 1-6. Psychoeducation will orient users to their upcoming experience, provide education about internalized weight bias, the chronic stress system, the utility of self-compassion practice to regulate physiological and psychological targets, and guidance on establishing, maintaining, and generalizing a mindfulness practice.
  Daily prompts: Participants will receive a text message every morning indicating their task for that day.
  Weekly prompts: Participants will receive a text message at the end of every week (Days 7, 14, 21, and 28) with a link to a brief adherence survey.
  Arms: Intervention

SUMMARY:
The proposed investigation is an experimental trial among 80 adults with obesity and internalized weight bias to determine preliminary effects of a smartphone-delivered brief self-compassion mindfulness intervention on internalized weight bias, compared to wait list control. All participants will receive a 4-week mindfulness-based intervention via smartphone. Participants will be randomly assigned to one of two treatment arms: (1) the intervention group, a self-compassion mindfulness practice tailored for weight and body concerns, or (2) a wait list control group, who will receive access to the intervention content following completion of end-of-treatment assessments. All intervention content will be delivered via text message.

DETAILED DESCRIPTION:
The proposed investigation is an experimental trial among 80 adults with obesity and internalized weight bias to determine preliminary effects of a smartphone-delivered brief self-compassion mindfulness intervention on internalized weight bias, compared to wait list control.

All participants will receive a 4-week mindfulness-based intervention via smartphone. Participants will be randomly assigned to one of two treatment arms: (1) the intervention group, a self-compassion mindfulness practice tailored for weight and body concerns, or (2) a wait list control group, who will receive access to the intervention content following completion of end-of-treatment assessments. All intervention content will be delivered via text message using Duke REDCap with Twilio integration. The intervention group will also complete psychoeducation on internalized weight bias and self-compassion. We will measure a number of potential moderating and mediating constructs, such as depression, trauma history, etc.

Intervention Components:

Intervention Group:

Guided Mindfulness Practice: Participants in the intervention group will receive compassion-based guided meditation audio recordings made publicly available by Kristin Neff at www.selfcompassion.org and Tara Brach at www.tarabrach.com. Many of these audio files were used in a previous investigation of self-compassion and body image (Albertson et al., 2015) and were selected due to their unique ability to target compassion and body concerns simultaneously. Daily mindfulness practice will require about 4-20 minutes per day to complete (days 2-28).

Psychoeducation: Participants in the intervention group will receive psychoeducation delivered via study website over days 1-6 (see Table 2). They will receive a new lesson via text message on each of these days, each covering a different topic related to the intervention. The purpose of the psychoeducation phase is to orient users to their upcoming experience, provide education about internalized weight bias, the chronic stress system, the utility of self-compassion practice to regulate physiological and psychological targets, and guidance on establishing, maintaining, and generalizing a mindfulness practice. Engagement in psychoeducation materials will take approximately 20-30 minutes per day (days 1-6).

Daily prompts: Participants will receive a text message every morning indicating their task for that day. Tasks include: review psychoeducation provided, or practice mindfulness today. Prompts will be brief and will require a minute or two to read. Assigned activity varies by day.

Weekly prompts: Participants will receive a text message at the end of every week (Days 7, 14, 21, and 28) with a link to a brief adherence survey. This will measure how many days they practiced that week. The brief adherence survey will take approximately 5 minutes to complete.

ELIGIBILITY:
Inclusion criteria:

* At least 18 years of age
* BMI at least 30 kg/m2
* Elevated weight bias internalization levels
* Must live within Eastern Standard Time zone
* Must own a smartphone and be willing to receive 1-2 text messages daily, practice mindfulness for approximately 20 minutes daily, and engage with weekly intervention content

Exclusion criteria:

* Under 18 years old
* BMI < 30
* No experienced or internalized weight bias reported
* Lives in another time zone (not EST)
* Currently attempting to lose weight or restrict diet
* Currently enrolled in an intervention for weight, weight bias, self-compassion or mindfulness
* Currently or recently a "regular meditator"
* Plans for bariatric surgery during or immediately following intervention period
* Investigator discretion for safety reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Change in Internalized Weight Bias | Baseline to End-of-treatment (4 weeks)
  Self-report measured using the Weight Bias Internalization Scale (WBIS-M)
Change in Weight Self-Stigma | Baseline to End-of-treatment (4 weeks)
  Self-report measured using the Weight Self-Stigma Questionnaire (WSSQ)
Change in Self-compassion | Baseline to End-of-treatment (4 weeks)
  Self-report measured using the Self Compassion Scale (SCS)

SECONDARY OUTCOMES:
Change in mindfulness | Baseline to End-of-treatment (4 weeks)
  Self-report measured using the Short-Form Five Facet Mindfulness Questionnaire (SF-FFMQ)

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Hopkins, MA, Principal Investigator — Duke University; Gary G Bennett, PhD, Principal Investigator — Duke University
Locations (1):
- Reuben-Cooke Building, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share de-identified study materials that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Materials will be available following completion of the trial and all planned publications.
Access Criteria: Individuals may request access to study materials for use in systematic reviews, metaanalyses, and other relevant uses. Please contact study PI (Hopkins) to request access.

REFERENCES:
- [Derived] Hopkins CM, Miller HN, Brooks TL, Mo-Hunter L, Steinberg DM, Bennett GG. Designing Ruby: Protocol for a 2-Arm, Brief, Digital Randomized Controlled Trial for Internalized Weight Bias. JMIR Res Protoc. 2021 Nov 25;10(11):e31307. doi: 10.2196/31307. PMID 34842549